CLINICAL TRIAL: NCT05036369
Title: A Prospective, Randomized, Multi-center, Double-Blinded, Clinical Study to Assess the Efficacy and Safety of Vibrant Capsule vs. Placebo, for the Treatment of Chronic Idiopathic Constipation
Brief Title: Vibrant Capsule vs. Placebo for Patient Suffering From Constipation
Acronym: Capsule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrant Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 280CLD
Record Dates: First submitted 2021-08-02; First posted 2021-09-05 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2023-07

CONDITIONS: Constipation Chronic Idiopathic
Keywords: Constipation; Vibrating capsule; Chronic Idiopathic Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: The objectives are to assess the efficacy and safety of Vibrant capsule administered twice a week
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study. The subjects and the evaluators will be blinded to the treatment allocated to each subject. Each site will assign an unblinded person that will handle all issues related to capsule administration and accountability. The unblinded person will not be involved in any subject's assessments. Rest of the site staff will remain blind throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active capsule (Experimental): The Vibrant non-biodegradable capsule administrated twice a week
  Interventions: Device: Vibrant capsule
- Placebo (Placebo Comparator): The placebo capsule is a softgel biodegradable capsule which is visually similar to the Vibrant active capsule and administrated twice a week
  Interventions: Device: Placebo capsule

INTERVENTIONS:
Device: Vibrant capsule — Vibrant capsule - Administered twice a week (Monday and Thursday).
  Arms: Active capsule
Device: Placebo capsule — Placebo Capsule administered twice a week (Monday and Thursday)
  Arms: Placebo

SUMMARY:
The objectives are to assess the efficacy and safety of Vibrant capsule administered twice a week

DETAILED DESCRIPTION:
The study is a prospective, randomized, multicenter, adaptive design, double blinded clinical study, to evaluate the efficacy and safety of Vibrant Capsule vs. placebo in relieving constipation in subjects with Chronic Idiopathic Constipation.

Two arms will be assessed (at a ratio of 1:1 of Vibrant Treatment vs. placebo):

* Vibrant Capsule administered twice a week (Monday and Thursday)
* Placebo Capsule administered twice a week (Monday and Thursday) Subjects will come for 4 visits: Screening (visit 1), baseline (visit 2), after 4 treatment weeks from baseline (visit 3) and after 8 treatment weeks from baseline (Final visit , visit 4). A total of 8 treatment weeks.

During the entire study period subjects will be asked to refrain from taking any medications or supplements to relieve their constipation.

Subjects will be authorized to use rescue medication after 3 consecutive days without a bowel movement

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 22 years and older
2. Subjects with Chronic Idiopathic Constipation (CIC) according to Rome IV criteria
3. Subjects who have not experienced relief of their symptoms from one or more available therapies (for at least one month at recommended dose) or unable to tolerate these therapies
4. Subjects with an average of ≤2.5 Spontaneous Bowel Movements (SBM) per week and ≥1 SBM per week (as a result of at least 1 SBM and not more than 3 SBMs during each of the run-in weeks)
5. Subjects above 50 years old or <50 years old and with alarm signs should have colonoscopy performed within 10 years prior to study participation. Colonoscopy results should exclude GI obstruction and/or GI malignancy
6. Subject signed the Informed Consent Form (ICF)
7. Female subjects must have a negative blood pregnancy test during screening, confirmed by a negative urine pregnancy test during baseline and must not be lactating prior to receiving study medication. For females of child-bearing potential, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. All other female subjects must have the reason for their inability to bear children documented in the medical record [i.e., tubal ligation, hysterectomy, or post-menopausal (defined as a minimum of one year since the last menstrual period)]; in these circumstances, a pregnancy test will not be necessary.

Exclusion Criteria:

1. History of complicated/obstructive diverticular disease
2. History of intestinal or colonic obstruction, or suspected intestinal obstruction.
3. History of significant gastrointestinal disorder, including any form of inflammatory bowel disease or gastrointestinal malignancy (celiac disease is accepted if the subject has been treated and is in remission)
4. Clinical evidence of current and significant gastroparesis
5. Use of any of the following medications:

   * Medications that may affect intestinal motility (including but not limited to prokinetics, anti-Parkinsonian medications, opiates, opioids, Verapamil, Nifedipine, iron, magnesium supplements, Tricyclic antidepressants (TCAs), Heparin, Warfarin and Baclofen.
   * With the exception of antidepressants (other than TCAs), thyroid or hormonal replacement therapy, when the subject has been on a stable dose for at least 3 months prior to enrollment.
6. Clinical evidence of significant respiratory, cardiovascular, renal, hepatic, biliary, endocrine, psychiatric or neurologic disease.
7. Presence of cardiac pacemaker, gastric electrical stimulator or any electrical implanted device.
8. History of, or current eating disorders, such as anorexia, bulimia, or compulsory overeating.
9. Diagnosis of mega-rectum or colon, congenital anorectal malformation, clinically significant rectocele, history of intestinal resection (with an exception for appendectomy, cholecystectomy and inguinal hernia repair), history of bariatric surgery or evidence of any structural abnormality of the gastrointestinal tract that might affect capsule's transit
10. History of Zenker's diverticulum, dysphagia, esophageal stricture, eosinophilic esophagitis or achalasia
11. Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs): chronic use is defined as taking full dose NSAIDs more than three times a week for at least six months. Subjects on cardiac doses of aspirin may be enrolled in the study
12. Subjects with pelvic floor dysfunction/defecatory disorder, based on subject history
13. Participation in another interventional clinical study within one month prior to screening.
14. Women who are pregnant or lactating
15. Use of any medication for constipation relief during the study, except as rescue medication, as indicated by study rules
16. Inability to use an electronic daily Diary (on a computer, phone application, tablet or other electronic device) to report bowel movements, symptoms and medication usage
17. Subject participated in a previous Vibrant study
18. Subjects planning to undergo MRI during the study
19. Any known allergy to soybean, beeswax, Calcium Carbonate, Gelatin, Glycerin or Titanium dioxide
20. Any other condition which in the opinion of the investigator may adversely affect the safety of the subject or would limit the subject's ability to complete the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tal Malina, MBA, Study Director — Vibrant Ltd.
Locations (2):
- United States (2):
  - Advanced Rx Clinical Research Group, Inc, Westminster, California
  - American Research Institute, INC, Cutler Bay, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruitment was conducted in 30 clinical sites in the USA from June 2021- September 2022
Pre-assignment Details: Following the consent process, subjects who met the study criteria started a run-in period of 2-4 weeks, during which they completed a daily eDiary with questions regrading their bowel movements and constipation symptoms.
Period: Overall Study
Arm/Group | Active Capsule | Placebo
Started | 44 | 56
Completed | 43 | 53
Not Completed | 1 | 3
Not completed — Run In non compliance | 1 | 2
Not completed — Change in eligibility criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Capsule | Placebo | Total
Number analyzed (Participants) | 44 | 56 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (12.87) | 41.8 (11.65) | 43.3 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 13 | 45
  Male | 12 | 43 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8 | 14 | 22
  Hispanic or Latino | 22 | 27 | 49
  Black or African American | 6 | 9 | 15
  Native American or American Indian | 1 | 1 | 2
  Asian/ Pacific Islander | 7 | 4 | 11
  Other | 0 | 1 | 1
Age of constipation onset (years) [Mean (Standard Deviation); unit: years] | 33.1 (13.80) | 29.6 (14.77) | 31.2 (14.39)

OUTCOME MEASURES:

1. Primary Outcome: CSBM 1 Success Rate
Description: CSBM1 Success Rate: defined as the number of Participants with an increase from the run-in period of at least one weekly Complete Spontaneous Bowel Movement (CSBM) during at least 6 of the 8 weeks of treatment.
  NOTE:
  A spontaneous bowel movement (SBM) is defined as a bowel movement that occurs at least 48h after laxative/rescue intake and without digital maneuver.
  A complete spontaneous bowel movement (CSBM) is defined as a spontaneous bowel movement associated with a feeling of complete evacuation by the subject.
Time Frame: up to 8 weeks of treatment
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Active Capsule | Placebo
Number analyzed (Participants) | 43 | 53
Participants | 24 | 17

2. Primary Outcome: CSBM2 Success Rate
Description: CSBM2 Success Rate: defined as the number of Participants with an increase from the run-in period of at least two weekly Complete Spontaneous Bowel Movement (CSBM) during at least 6 of the 8 weeks of treatment.
  NOTE:
  A spontaneous bowel movement (SBM) is defined as a bowel movement that occurs at least 48h after laxative/rescue intake and without digital maneuver.
  A complete spontaneous bowel movement (CSBM) is defined as a spontaneous bowel movement associated with a feeling of complete evacuation by the subject.
Time Frame: up to 8 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Active Capsule | Placebo
Number analyzed (Participants) | 43 | 53
Participants | 13 | 12

3. Secondary Outcome: Straining Based on the Subject's Assessment Recorded in Daily Diaries
Description: Change from baseline in average straining based on the subject's account in daily diary reports.
  The straining level reported by the patient on a scale ranged from 0 - No straining to 10 Unbearable straining.
Time Frame: up to 10 weeks
Population: mITT
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Capsule | Placebo
Number analyzed (Participants) | 43 | 53
units on a scale | -2.4 [-3.14 to -1.66] | -1.70 [-2.31 to -1.08]

4. Secondary Outcome: CSBM1 Expanded Success Rate,
Description: CSBM1 expanded success rate, defined as the number of Participants with an increase from the run-in period of at least one weekly Complete Spontaneous Bowel Movement (CSBM) during at least 5 of the 8 weeks of treatment.
Time Frame: up to 8 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Active Capsule | Placebo
Number analyzed (Participants) | 43 | 53
Participants | 28 | 23

5. Secondary Outcome: CSBM2 Expanded Success Rate
Description: defined as the number of Participants with an increase from the run-in period of at least two weekly Complete Spontaneous Bowel Movement (CSBM) during at least 5 of the 8 weeks of treatment.
Time Frame: up to 8 weeks of treatment
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Active Capsule | Placebo
Number analyzed (Participants) | 43 | 53
Participants | 14 | 14

6. Secondary Outcome: Change From Baseline in Stool Consistency
Description: Change from baseline in average stool consistency, using the Bristol Stool Scale (1-7) where 1 = Separate hard lumps, like nuts (hard to pass) and 7 =watery, no solid pieces, entirely liquid
Time Frame: up to 10 weeks
Population: mITT
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Capsule | Placebo
Number analyzed (Participants) | 43 | 53
units on a scale | 1.31 [0.84 to 1.78] | 0.81 [0.42 to 1.20]

ADVERSE EVENTS:
Time Frame: The Safety reporting conducted throughout the treatment period (8 weeks)
Arm/Group | Active Capsule | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/44 | 1/56
Other Adverse Events (participants affected / at risk) | 16/44 | 11/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Capsule (N=44) | Placebo (N=56)
Hospitalized due to bleeding from the catheter port (Renal and urinary disorders) | 0 (0) | 1 (1) — Hospitalized due to bleeding from the catheter port
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Capsule (N=44) | Placebo (N=56)
Headache (Nervous system disorders) | 3 | 1
Sensation of Vibration (Product Issues) | 7 | 0
Heartburn (Gastrointestinal disorders) | 1 | 0 — Heartburn
UTI (Renal and urinary disorders) | 1 | 0 — Urinary tract infections
Diarrhea (Gastrointestinal disorders) | 1 | 0 — Diarrhea
Vomiting (Gastrointestinal disorders) | 0 | 1 — Vomiting
Fatigue (General disorders) | 0 | 1 — Fatigue
Esophageal Spasm (Gastrointestinal disorders) | 0 | 1 — Esophageal Spasm
Nausea (Gastrointestinal disorders) | 0 | 1 — Nausea
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 — Gastroenteritis
Other (General disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Permission to use study data is required

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT05036369/Prot_SAP_001.pdf